CLINICAL TRIAL: NCT06951087
Title: Effect of Intravitreal and Intracameral Injection of Dexamethasone Sodium Phosphate on Mild to Moderate NPDR During Cataract Phacoemulsification
Brief Title: Intravitreal and Intracameral DEX in NPDR
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-K068; 81974129, 82171038, 82101101 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2025-01-07; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-12

CONDITIONS: Non-Proliferative Diabetic Retinopathy
Keywords: non-proliferative diabetic retinopathy; cataract phacoemulsification; cystoid macular edema
MeSH Terms: conditions — Macular Edema | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intravitreal DEX group (Experimental): Patients received an intravitreal injection of 0.5 mg DEX during phacoemulsification in the intravitreal DEX group
  Interventions: Drug: Dexamethasone sodium phosphate
- intracameral DEX group (Experimental): Patients received an intracameral injection of 0.5 mg DEX during phacoemulsification in the intracameral DEX group
  Interventions: Drug: Dexamethasone sodium phosphate
- the control group (No Intervention): Patients received no injection during phacoemulsification in the control group

INTERVENTIONS:
Drug: Dexamethasone sodium phosphate — In patients with stable DR and no significant macular edema, intravitreal anti-VEGF injections after phacoemulsification surgery can prevent the worsening of postoperative macular edema and potentially improve final visual outcomes while maintaining safety. Laser coagulation and intravitreal anti-VEGF injections are currently considered the standard treatments for PDR. However, the cost of anti-VEGF drugs often prevents many patients from receiving regular and timely injections. Intravitreal corticosteroids may be used as an alternative to anti-VEGF agents.
  Arms: intracameral DEX group; intravitreal DEX group

SUMMARY:
To investigate the effects of intravitreal and intracameral injection of dexamethasone during cataract phacoemulsification in patients with mild to moderate non-proliferative diabetic retinopathy

DETAILED DESCRIPTION:
The study aims to analyze the impact of intravitreal and intracameral DEX in diabetic patients with NPDR who are undergoing phacoemulsification surgery. Specifically, the investigators will investigate its effects on postoperative macular central thickness, the development of DME, and the progression of DR.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetic cataracts patients who were diagnosed with mild to moderate NPDR

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
measure the central point thickness (CPT) and central foveal thickness (CFT) | From enrollment to the end of treatment at 3 months
  optical coherence tomography (OCT) was used to perform the retinal examination, macular cube scans (512 × 128) and measure the central point thickness (CPT) and central foveal thickness (CFT). The CPT measurement focused on a central circle with a diameter of 1mm, and the CFT was calculated as the average of three consecutive measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute, Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes